CLINICAL TRIAL: NCT03093350
Title: Tumor Associated Antigen (TAA) Specific Cytotoxic T Lymphocytes Administered in Patients With Breast Cancer
Brief Title: TACTIC - TAA Specific Cytotoxic T Lymphocytes in Patients With Breast Cancer
Acronym: TACTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); National Cancer Institute (NCI) (NIH); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-39209 TACTIC; P50CA186784 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tumor Associated Antigen Specific T cells
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAA-Specific CTLs (Experimental): Patients receiving TAA-specific CTLs as therapy for breast cancer.
  Interventions: Biological: TAA-specific CTLs

INTERVENTIONS:
Biological: TAA-specific CTLs — Each patient will receive 2 injections at a fixed dose, 28 days apart, according to the following dose schedule: The expected volume of infusion will be 1 to 10 cc.
  Dose schedule:
  Day 0: 2 x 10^7 cells/m2
  Day 28: 2 x 10^7 cells/m2
  If patients have stable disease or a partial response by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria at their 6 week evaluation after the 2nd cell dose, they will be eligible to receive up to 6 additional doses of CTLs, At least one month should have passed before each additional dose.. Each additional infusion will consist of the same cell number or less (if there is not enough product available for the subject's original dose) than their second infusion. Patients will not be able to receive additional doses until the initial safety profile is completed at 6 weeks following the second infusion.

SUMMARY:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

The study is being conducted in patients in which breast cancer has come back after standard treatment. Volunteers in this research study are treated using special immune system cells called tumor-associated antigen (TAA)-specific cytotoxic T lymphocytes, a new experimental therapy.

The proteins that investigators are targeting in this study are called tumor-associated antigens (TAAs). These are cell proteins that are specific to the cancer cell. They do not show, or they show up in low quantities, on normal human cells. In this study, investigators target five common TAAs. They are called NY-ESO-1, MAGEA4, PRAME, Survivin and SSX2. On a different study, patients have been treated and so far this treatment has shown to be safe.

Investigators now want to try this treatment in patients with breast cancer.

These TAA-specific cytotoxic T lymphocytes (TAA-CTLs) are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to determine the clinical efficacy of TAA-specific CTLs, to learn what the side-effects are, and to see whether this therapy might help patients with breast cancer.

DETAILED DESCRIPTION:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

Investigators will take a maximum of approximately 79 teaspoons of blood from patients on one to three occasions over a two-month period. Under certain conditions related to the patient's health, blood may be collected using a process called apheresis. Apheresis is the process where blood is passed through a machine that separates out the components of blood that we need. The remainder of the patient's blood will then be returned to his/her body.

Investigators will use this blood to grow T cells. Investigators will first grow a special type of cells called dendritic cells which will activate T cells. Once these are made, investigators will load them with small pieces of protein called peptides taken from the TAAs that we want to target. This helps train the T cells to kill cancer cells which express TAAs on their surface. Then the TAA-specific CTLs are expanded.

The cells will be infused by intravenous infusion (IV) into the patient over 1-10 minutes. The patient may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Acetaminophen (Tylenol) and diphenhydramine (Benadryl) are given to prevent a possible allergic reaction to the TAA-CTL administration. Initially, two doses of TAA-CTLs will be given four weeks apart. The patient's cancer will be assessed pre-infusion, and then 6 weeks after the second infusion. If after the second infusion there is a reduction in the size of the patient's tumor on Computed Tomography (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET) as assessed by a radiologist, the patient can receive up to six (6) additional doses of the TAA-CTLs if they wish. At least one month should pass before each additional dose. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

In between the first and second TAA-CTL infusions, and for 6 weeks after the 2nd infusion, the patient should not receive any other anti-cancer treatments such as radiation therapy or chemotherapy. If the patient does receive any other therapies in-between the first and second infusion of TAA-CTLs, they will be taken off treatment and will not be able to receive the second infusion.

MEDICAL TESTS BEFORE TREATMENT:

Before being treated, patients will receive a series of standard medical tests:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurements of the patient's tumor by routine imaging studies.
* Pregnancy test if the patient is a female who can have children.

MEDICAL TESTS DURING TREATMENT:

Patients will receive standard medical tests on the day of their second and subsequent infusions:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function.

MEDICAL TESTS AFTER TREATMENT

- Imaging study 6 weeks after the 2nd TAA-CTL infusion.

To learn more about the way the TAA-CTLs are working in the patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each infusion, at Weeks 1, 2, and 4 after the first cell dose and at Weeks 1, 2, 4 and 6 after the second cell dose. Afterwards, blood will be collected at 3, 6, 9 and 12 months after the 2nd infusion. Investigators will use this blood to see how long the TAA-CTLs last, and to look at the patient's immune system response to the cancer. The immune system is part of the body that helps protect against disease.

Study Duration: The patient's active participation in this study will last for approximately one (1) year. If the patient receives additional doses of the TAA-CTLs as described above, his/her active participation will last until one (1) year after the last dose. Investigators will then contact the patient once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate the patient's disease response long-term.

ELIGIBILITY:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

PROCUREMENT INCLUSION CRITERIA:

1. Any breast cancer patient with metastatic or locally recurrent unresectable disease.
2. Patients with life expectancy greater than or equal to 12 weeks.
3. Age greater than or equal to 18 and less than or equal to 80 years old.
4. Hgb greater than or equal to 7.0.
5. Informed Consent explained to, understood by and signed by patient. Patient given copy of informed consent.

TREATMENT INCLUSION CRITERIA:

1. Any breast cancer patient with metastatic or locally recurrent unresectable breast cancer currently progressive, after at least two prior lines of therapy in the advanced setting. Patients with HER2+ disease must have failed two or more different anti-HER2 agents.
2. Patients must have measurable or evaluable disease per RECIST 1.1 criteria.
3. Patients with life expectancy greater than or equal to 12 weeks.
4. Age greater than or equal to 18 and less than or equal to 80 years old.
5. Pulse oximetry of greater than 95% on room air.
6. Patients with ECOG score less than or equal to 2 or a Karnofsky score of greater than or equal to 50.
7. Patients with bilirubin less than or equal to 2x upper limit of normal, AST less than or equal to 3x upper limit of normal, and Hgb greater than or equal to 7.0.
8. Patients with a creatinine normal for age.
9. Patients should have been off other investigational therapy for one month prior to receiving treatment on this study.
10. Patients should have been off conventional therapy for at least 1 week prior to receiving treatment on this study.
11. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the T cell infusion.
12. Informed Consent explained to, understood by and signed by patient. Patient given copy of informed consent.

PROCUREMENT EXCLUSION CRITERIA:

1. Patients with severe intercurrent infection.
2. Patients with active HIV infection at time of procurement.
3. Patients with a chronic uncontrolled medical condition that, in the opinion of the principal investigator, precludes them from participation.

TREATMENT EXCLUSION CRITERIA:

1. Patients with severe intercurrent infection.
2. Patients receiving systemic corticosteroids (Patients off steroids for at least 48 hours are eligible).
3. Pregnant or lactating.
4. Patients with a chronic uncontrolled medical condition that, in the opinion of the principal investigator, precludes them from participation.
5. HIV positive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar F Rimawi, MD, Principal Investigator — Baylor College of Medicine; Anne Leen, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Smith Clinic - Harris Health System, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TAA-Specific CTLs: Patients receiving TAA-specific CTLs as therapy for breast cancer.
  TAA-specific CTLs: Each patient will receive 2 injections at a fixed dose, 28 days apart, according to the following dose schedule: The expected volume of infusion will be 1 to 10 cc.
  Dose schedule:
  Day 0: 2 x 10^7 cells/m2
  Day 28: 2 x 10^7 cells/m2
  If patients have stable disease or a partial response by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria at their 6 week evaluation after the 2nd cell dose, they will be eligible to receive up to 6 additional doses of CTLs, At least one month should have passed before each additional dose.. Each additional infusion will consist of the same cell number or less (if there is not enough product available for the subject's original dose) than their second infusion. Patients will not be able to receive additional doses until the initial safety profile is completed at 6 weeks following the second infusion.
Period: Overall Study
Arm/Group | TAA-Specific CTLs
Started | 12
Started Treatment | 10
Completed | 10
Not Completed | 2
Not completed — Death | 1
Not completed — Signed consent, never began treartment | 1

BASELINE CHARACTERISTICS:
Population: 12 patients were enrolled, but 10 were assigned to treatment. 1 patient signed consent but never began treatment, and 1 patient died before treatment began.
Arm/Group | TAA-Specific CTLs
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.80 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Evaluable Patients With Complete Response or Partial Response or Stable Disease for ≥10 Weeks From the First Infusion (6 Weeks After the Second Infusion) According to the RECIST Criteria
Description: To determine the clinical efficacy associated with the administration of multiTAA-specific T cells in breast cancer patients with metastatic or locally recurrent unresectable disease as measured by clinical benefit rate (defined as overall response plus stable disease for 10 weeks or longer). Per the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria and assessed by CT or MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter (LD) of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; Overall Response (OR) = CR + PR.
Time Frame: 12 weeks
Population: 12 patients were enrolled, but 10 were assigned to treatment. 1 patient signed consent but never began treatment, and 1 patient died before treatment began. 9 patients completed treatment; 1 patient progressed prior to 2nd infusion and was considered inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | TAA-Specific CTLs
Number analyzed (Participants) | 9
Participants | 1

2. Secondary Outcome: Median Progression-free Survival
Description: To evaluate the progression-free survival of patients after multiTAA-specific T cell infusion. Progression is defined, according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Criteria, as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 1 year
Population: 12 patients were enrolled, but 10 were assigned to, and began, treatment. 1 patient signed consent but never began treatment, and 1 patient died before treatment began.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TAA-Specific CTLs
Number analyzed (Participants) | 10
days | 69.5 [13 to 72]

3. Secondary Outcome: Median Overall Survival
Description: To evaluate the overall survival of patients after multiTAA-specific T cell infusion
Time Frame: 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TAA-Specific CTLs
Number analyzed (Participants) | 10
days | 116 [37 to NA] — Not enough participants had event to calculate upper 95% CI.

ADVERSE EVENTS:
Time Frame: 10 weeks (from date of 1st injection up to 6 weeks after date of 2nd injection) for adverse events, and 1 year (from date of 1st injection) for all-cause mortality.
Description: Adverse events were assessed starting at the date of 1st injection, then at 1 week after 1st injection, 2 weeks after 1st injection, date of 2nd injection (4 weeks after 1st injection), 1 week after 2nd injection, 2 weeks after 2nd injection, 4 weeks after 2nd injection, and 6 weeks after 2nd injection using descriptions and grading scales found in CTCAE v4.0. All-cause mortality was assessed for 1 year from the date of 1st injection.
Arm/Group | TAA-Specific CTLs
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAA-Specific CTLs (N=10)
Fever (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAA-Specific CTLs (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03093350/Prot_SAP_000.pdf